CLINICAL TRIAL: NCT04709289
Title: Adverse Effects of ALA-PDT for the Treatment of Moderate to Severe Acne
Brief Title: Adverse Effects of ALA-PDT for the Treatment of Moderate to Severe Acne Vulgaris: a Prospective Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Dermatology Hospital (Other)
Responsible Party: Principal Investigator, Xiuli Wang, Director, Clinical Professor, Shanghai Dermatology Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-04
Record Dates: First submitted 2021-01-10; First posted 2021-01-14 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Aminolevulinic Acid; Photochemotherapy

STUDY DESIGN:
Masking Description: Evaluator assesses photographs without prior knowledge of intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Conventional Photodynamic Therapy(C-PDT) group (Experimental): The conventional photodynamic therapy(C-PDT) group underwent narrow-band light-emitting diode (LED) irradiation (630 nm; 140 J/cm2) after applying 5% 5-aminolevulinic acid cream for 3h.A repeat treatment was administered once every two weeks for 3 times.
  Interventions: Other: Aminolevulinic acid, photodynamic therapy

INTERVENTIONS:
Other: Aminolevulinic acid, photodynamic therapy — Aminolevulinic acid, photodynamic therapy

SUMMARY:
To understand, prevent and treat the adverse reactions more comprehensively, we sought to systemically document the adverse effects of ALA-PDT for moderate to severe acne vulgaris.

DETAILED DESCRIPTION:
To understand, prevent and treat the adverse reactions more comprehensively, we sought to systemically document the adverse effects of ALA-PDT for moderate to severe acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* (1) Patients diagnosed with moderate to severe acne and graded grade III-IV according to Investigator's Global Assessment (IGA) ;
* (2) Patients unsuitable for drug treatment owing to various reasons and who voluntarily participated and signed informed consent following information about other alternatives;
* (3) Patients who read the instructions and were willing to follow the program requirements.

Exclusion Criteria:

* (1) Patients who had a history of photosensitive diseases;
* (2) Patients who had Modified-PDT;
* (3) Patients who had oral isotretinoin in the past 3 months, used oral contraceptives or antibiotics and underwent local or facial surgery in the past 4 weeks;
* (4) Female patients who were pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
The clearance rate of lesions | 1 week after treatment
  The change rate in lesion clearance of acne vulgaris at 7 days after treatment will be measured as the primary outcome

SECONDARY OUTCOMES:
Assessment of adverse effects | up to 7 days after treatment.
  the incidence, severity, occurrence and duration time of erythema, pain, burning skin, itching, pustule, exudation, edema, blister, dry skin, crust and hyperpigmentation of last treatment, as well as lesion photos were detailed asked and recorded during the clinical encounter, up to 7 days after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Xiuli Wang, MD PhD, Study Director — Shanghai Skin Disease Hospital
Locations (1):
- Lei Shi, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes